CLINICAL TRIAL: NCT01963715
Title: A Phase 1, Multi-center, Open-label Study of IMGN289 Administered Intravenously in Adult Patients With EGFR-positive Solid Tumors
Brief Title: A Phase 1 Study of IMGN289 in Adult Patients With EGFR-positive Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMGN0501
Record Dates: First submitted 2013-10-09; First posted 2013-10-16 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: EGFR Positive Solid Tumors
Keywords: IMGN289; Antibody Drug Conjugate; antibody; EGFR; NSCLC; SCCHN; Head and neck; Squamous cell carcinoma; Solid tumor; Immunogen; Lung; Phase 1
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EGFR+ Solid Tumor (Experimental): EGFR+ Solid Tumor
  Interventions: Drug: IMGN289

INTERVENTIONS:
Drug: IMGN289

SUMMARY:
This is a Phase 1, first-in-human study to determine the recommended dose of IMGN289 in adult patients with advanced EGFR-positive tumors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old at time of consent
* Diagnosed with a solid tumor that has progressed despite standard therapy or for which no standard effective or curative options exist or are suitable
* EGFR-positive tumor expression
* Adequate blood and organ function
* Must agree to use contraception while on study and for 12 weeks after the last dose of IMGN289 as applicable
* Must be willing and able to sign informed consent and follow the study schedule and other protocol requirements

Exclusion Criteria:

* Other anti-cancer treatment during the study
* Symptomatic brain metastases
* Other clinically significant disease as defined by the protocol
* Chronic skin condition that requires prescribed oral or intravenous treatment
* History of severe rash that required discontinuation of prior EGFR targeted therapy
* Receiving therapeutic doses of warfarin or heparin for anti-coagulation
* Known diagnosis of HIV or active viral hepatitis
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | Up to 2 years

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 2 years
Area under the plasma concentration versus time curve | Up to 2 years
  Determine the amount of IMGN289 in participants blood (pharmacokinetics)
Peak plasma concentration (Cmax) of IMGN289 | Up to 2 years
  Determine the amount of IMGN289 in participants blood (pharmacokinetics)
Presence of Human Anti Human Antibody and Human Anti Drug Antibody | Up to 2 years
  Assess whether participants develop an immune response to IMGN289
Tumor measurements per RECIST 1:1 | Up to 2 years
  Assess preliminary anti-tumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vergara-Silva, MD, Study Director — ImmunoGen, Inc.
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan